CLINICAL TRIAL: NCT06974344
Title: Randomized Controlled Trial Protocol Comparing Splenic Artery Ligation Versus Octreotide for Portal Flow Modulation (SCALOP) in Living Donor Liver Transplantation
Brief Title: Octreotide vs. Splenic Artery Ligation for Portal Flow Modulation in Living Donor Liver Transplants (SCALOP Trial)
Acronym: SCALOP
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: King Faisal Specialist Hospital & Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RAC2241241
Record Dates: First submitted 2025-04-15; First posted 2025-05-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-04

CONDITIONS: Small-for-Size Syndrome
Keywords: Living Donor Liver Transplantation; LDLT; Small-for-Size Graft; SFS; Portal Flow Modulation; Graft Inflow Modulation; Octreotide; Somatostatin Analogue; Splenic Artery Ligation,; SAL; Randomized Controlled Trial; RCT; Complications; Outcomes; Mortality; Liver Hemodynamics; Early Allograft Dysfunction; Small-for-Size Syndrome; SFSS; Survival
MeSH Terms: interventions — Octreotide; Pharmaceutical Preparations

STUDY DESIGN:
Intervention Model Description: This is a parallel-group, randomized, single-blind trial comparing octreotide infusion versus splenic artery ligation for portal flow modulation in living donor liver transplantation. While participants are initially assigned to one treatment arm, crossover to the alternative therapy is permitted as rescue treatment if hemodynamic targets are not met. Outcome assessors will remain blinded to the original allocation throughout follow-up.
Who Masked: Participant, Outcomes Assessor
Masking Description: Biostatistician
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Octreotide Infusion Arm (Active Comparator): Continuous intravenous octreotide (1 mcg/kg/hr) initiated at liver graft reperfusion and continued postoperatively until hemodynamic stability is achieved.
  Interventions: Drug: Octreotide (drug)
- Splenic Artery Ligation (SAL) Arm (Active Comparator): Intraoperative ligation of the splenic artery using non-absorbable suture near its origin.
  Interventions: Procedure: Splenic Artery Ligation (SAL)

INTERVENTIONS:
Drug: Octreotide (drug) — Continuous intravenous octreotide acetate infusion initiated at hepatic reperfusion during living donor liver transplantation (LDLT). The initial dose is 1 mcg/kg/hr, titrated intraoperatively based on portal venous flow (PVF) and hepatic artery flow / resistive index (RI) measurements. The infusion continues postoperatively in the ICU until stable graft hemodynamics are achieved (target PVF <5 mL/min/g and presence of diastolic hepatic arterial flow). Dose adjustments are permitted for efficacy or safety concerns, with all modifications documented. The intervention is administered via central venous access using standard infusion protocols
  Other Names: Octreotide acetate; Sandostatin®; Somatostatin analogue
  Arms: Octreotide Infusion Arm
Procedure: Splenic Artery Ligation (SAL) — Intraoperative ligation of the splenic artery performed during living donor liver transplantation (LDLT) using non-absorbable suture material (e.g., polypropylene). The ligation is typically placed near the splenic artery origin for maximal portal flow modulation, with exact positioning determined by surgeon assessment of vascular anatomy and intraoperative hemodynamics (targeting portal venous flow <5 mL/min/g). The procedure is performed under direct visualization during the transplant operation, with post-ligation Doppler ultrasound confirmation of hemodynamic response within 60 minutes of biliary anastomosis.
  Arms: Splenic Artery Ligation (SAL) Arm

SUMMARY:
The goal of this clinical trial is to compare two treatments for regulating blood flow in small liver grafts during living donor liver transplantation (LDLT). The main questions it aims to answer are:

* Is octreotide (a medication) as effective or better than splenic artery ligation (surgery) in reducing complications after transplantation?
* Which treatment better controls blood flow while causing fewer side effects?

Researchers will compare octreotide (given through an IV) to splenic artery ligation (performed during surgery) to see which approach works best for patients receiving small liver grafts.

Participants will:

* Be randomly assigned to receive either octreotide or splenic artery ligation during their transplant surgery
* Have their liver blood flow monitored closely during and after surgery

Be followed for 90 days and 1 year to track complications, hospital stay, recovery, and survival.

This study may help doctors choose safer, more effective treatments for patients needing small liver grafts.

DETAILED DESCRIPTION:
This randomized controlled trial (SCALOP-RCT) investigates two strategies for managing portal hyperperfusion in adults receiving small living donor liver transplants (graft-to-recipient weight ratio <0.80%). Small grafts are prone to injury from high venous portal and low hepatic artery flow, leading to small-for-size syndrome (SFSS), a major cause of transplant failure.

Interventions Compared

* Octreotide: A somatostatic analogue that reduces portal venous flow and increased hepatic artery flow to the liver by constricting blood vessels, given continuously through an IV during and after surgery.
* Splenic Artery Ligation (SAL): A surgical procedure that ties off the artery supplying the spleen, indirectly lowering portal venous flow.

Study Design

* Randomization: Participants are assigned 1:1 to octreotide or SAL during transplant surgery.
* Rescue Protocol: If portal venous flow remains too high after the initial treatment, patients may switch to the alternative therapy (crossover).
* Blinding: Surgeons know the treatment, but outcome assessors and data analysts do not.

Key Assessments

* Primary: Total complication burden at 90 days (Comprehensive Complication Index(R) (CCI(R)).
* Secondary: Blood flow measurements, early liver function, hospital stay, survival, and quality of life.
* Rationale: Current approaches vary widely, with no consensus on whether medications or surgery work better. This trial will provide evidence to standardize care, potentially improving graft survival and expanding donor options.
* Population: 80 adults (18-70 years) undergoing LDLT at a single tertiary center.
* Innovation: First head-to-head comparison of these strategies with rigorous hemodynamic monitoring and crossover rescue design.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 and <70 years
2. Male and female genders
3. Undergoing Living Donor Liver Transplant (LDLT)
4. All indications
5. Receiving a small-for-size graft requiring portal flow modulation
6. Informed consent provided.

Exclusion Criteria:

1. Deceased Donor Liver Transplantation (DDLT)
2. Dual LDLT or dual LDLT/DDLT
3. Pregnancy
4. Known allergy to Octreotide / Somatostatin analogue

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2030-05-01 (Estimated); Study Completion 2030-09-01 (Estimated)

PRIMARY OUTCOMES:
Median Comprehensive Complication Index® (CCI®) | From the day of liver transplantation (Day 0) through postoperative day 90.
  The Comprehensive Complication Index® (CCI®) is a validated, quantitative metric that reflects the cumulative burden of postoperative complications by integrating all complications experienced by a patient into a single continuous scale (range: 0 (no complications) to 100 (death)). The CCI® is calculated using the Clavien-Dindo Classification to grade the severity of each complication (Grades I-V), with weights assigned based on clinical impact.
Small-for-size syndrome (SFSS) rate | From the day of liver transplantation (Day 0) through postoperative day 14
  SFSS is a clinically defined syndrome occurring in recipients of small-for-size liver grafts (graft-to-recipient weight ratio (GRWR) <0.80%), characterized by:
  * Persistent cholestasis (serum total bilirubin >5.8 mg/dL beyond postoperative day 14)
  * Refractory ascites (daily ascitic fluid output >1 L despite diuretics beyond day 14)
  * Coagulopathy (INR >2 with hypoalbuminemia <2.5 g/dL beyond day 14)
  Diagnostic Criteria
  * Requires ≥2 of the above features (per ILTS-iLDLT-LTSI 2023 Consensus Guidelines).
  * Excludes other causes of graft dysfunction (e.g., hepatic artery thrombosis, acute rejection).
Number and proportion of postoperative complication types and grades within 90 days | From the day of liver transplantation (Day 0) through postoperative day 90
  All complications occurring within 90 days post-transplantation will be prospectively recorded and graded using the Clavien-Dindo Classification, a validated system for surgical morbidity.
  * Grade I: Minor deviations (e.g., antipyretics for fever, bedside wound care).
  * Grade II: Pharmacological treatment (e.g., antibiotics for infection).
  * Grade III: Surgical/endoscopic intervention (IIIa: local anesthesia; IIIb: general anesthesia).
  * Grade IV: Life-threatening (IVa: single-organ dysfunction; IVb: multi-organ failure).
  * Grade V: Death.
Adequate portal flow modulation response rate | From intervention completion (T=0) to 60 minutes post-intervention
  The proportion of patients achieving target hemodynamic parameters following intervention (octreotide or splenic artery ligation), defined as:
  * Portal venous flow (PVF) <5 mL/min/graft weight and
  * Presence of diastolic hepatic arterial flow on Doppler ultrasound post-intervention.
Mortality rate | From the day of liver transplantation (Day 0) through postoperative day 90
  All-cause mortality occurring within 90 days post-transplantation, regardless of relationship to the intervention or underlying liver disease. This will the proportion of deaths over total number of patients within each arm and reported in percentage.

SECONDARY OUTCOMES:
Median portal venous flow (PVF) rate on intraoperative Liver Doppler ultrasound | Intraoperative (post-reperfusion) and postoperative (daily) timepoints until day 20 postoperatively or hospital discharge
  Portal venous flow (PVF): Volume flow rate (mL/min) normalized to graft weight (mL/min/g)
Median Hepatic artery resistive index (RI) on intraoperative Liver Doppler ultrasound | Intraoperative (post-reperfusion) and postoperative (daily) timepoints until day 20 postoperatively or hospital discharge
  Hepatic artery resistive index (RI): (Peak systolic velocity - End diastolic velocity)
Hepatic artery diastolic flow rate | Intraoperative (post-reperfusion) and postoperative (daily) timepoints until day 20 postoperatively or hospital discharge
  Binary presence or absence rate of end- diastolic flow on Liver Doppler Ultrasound
Median intensive care unit length of stay in days | Days from admission to the Intensive Care Unit (ICU) (typically Day 0 to Day 4 postoperatively) until ICU discharge to the surgical ward.
  Total number of days in the Intensive care unit (ICU) during the primary admission, from the day of transplant (Day 0) until discharge to the surgical ward.
Median hospital length of stay in days | From the day of liver transplantation (Day 0) until hospital discharge (typically day 20 postoperatively)
  Total number of days patient hospitalized during the index procedure
Graft survival rate at 1-year post-transplantation | From the day of liver transplantation (Day 0) through postoperative day 365
  The proportion of patients with a functional liver graft (alive without retransplantation) at 1 year post-transplant, analyzed by including all graft losses (death or retransplantation) using the Kaplan-Meier test.
Patient survival rate at 1-year post-transplantation | From the day of liver transplantation (Day 0) through postoperative day 365
  The proportion of patients with alive at 1 year post-transplant, analyzed using the Kaplan-Meier test.
Quality of Life Assessment (36-Item Short Form Health Survey, SF-36) (median values) | Measured at baseline (pre-transplant), 3 months, 6 months, and 12 months post-transplantation.
  The 36-Item Short Form Health Survey (SF-36) is a validated patient-reported outcome measure that assesses health-related quality of life. The SF-36 consists of eight subscales, which are further summarized into two component scores:
  * Physical Component Summary (PCS): Includes physical functioning, role-physical, bodily pain, and general health.
  * Mental Component Summary (MCS): Includes vitality, social functioning, role-emotional, and mental health.
  Scoring: Each subscale is scored from 0 to 100, where higher scores indicate better health-related quality of life. The median scores will be compared between the two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Dieter C. Broering, MD, PhD, Principal Investigator — Organ Transplant Center of Excellence, King Faisal Specialist Hospital and Research Center, Riyadh, Saudi Arabia; Dimitri A. Raptis, MD, MSc, PhD, Principal Investigator — Organ Transplant Center of Excellence, King Faisal Specialist Hospital and Research Center, Riyadh, Saudi Arabia; Massimo Malago, MD, PhD, Principal Investigator — Organ Transplant Center of Excellence, King Faisal Specialist Hospital and Research Center, Riyadh, Saudi Arabia
Locations (1):
- Organ Transplant Center of Excellence, King Faisal Specialist Hospital and Research Center, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data will be made available, including baseline demographic and clinical characteristics, detailed intervention parameters, outcome measures , and adverse event records. Supporting study documents including the final study protocol, statistical analysis plan, case report forms, and clinical study report synopsis will be shared to facilitate interpretation. These data will become accessible 12 months after publication of the primary study findings and remain available for ten years through a secure data repository.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Start date: Publication of the study. End date: One year after publication of the study
Access Criteria: Qualified researchers may request access by submitting a methodologically sound proposal for approval by the Principal Investigators and Data Monitoring Committee.